## Statistical Analysis Plan

**Official Title:** Motivational Enhancement to Augment Contingency Management for SARS-CoV-2 Testing and Vaccination Utilization Among Syringe Exchange Clients

NCT number: NCT05534061 Document Date: July 26, 2022

## Statistical Analysis Plan

Study Title: Creating a Sustainable Infrastructure for SARS-COV-2 Testing at Syringe Exchange

Programs

**Protocol Number:** 11162020.013

Preliminary analyses included a description of the sample and extent of missing data and tests of baseline equivalency of randomized groups. Study participants received the intervention across nine sites resulting in a multilevel data structure. We used multilevel logistic regression estimated with the generalized linear model using the adaptive quadrature quasi-likelihood estimator to compare rates of COVID-19 testing and vaccination administered on the same day of the intervention and anytime during the 9-month follow-up period. A Bernoulli distribution and logit link function were specified, and odds ratios and 95% confidence intervals reported to facilitate interpretation. First, a null model was specified to estimate the variability between sites and within individuals followed by the full model that included the study randomized condition as the predictor (coded 1 = CM + Connect2Test, 0 = CM).